CLINICAL TRIAL: NCT00561197
Title: An Open-label, Single-center, Phase 1/ 2 Study of Chemoradiotherapy and AT-101 in Patients With Locally Advanced Esophageal or Gastroesophageal Junction Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Drug not being developed for this indication
Sponsor: Ascenta Therapeutics (Industry)
Responsible Party: Kimberli Brill, Associate Director, Clinical Development, Ascenta Therapeutics
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AT-101-CS-102
Record Dates: First submitted 2007-11-19; First posted 2007-11-20 (Estimated); Last update posted 2013-01-04 (Estimated); Status verified 2013-01

CONDITIONS: Locally Advanced Esophageal or GE Junction Cancer
MeSH Terms: interventions — gossypol acetic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: AT-101 — Patients will receive AT-101 starting at 10 mg once daily for 5 of 7 days in conjunction with RT (50.4 Gy for 28 fractions) for approximately 5.5 weeks. Concurrently, patients will receive docetaxel (20 mg/m2) IV weekly (Monday) and 5-fluorouracil (300 mg/m2) as a 24 hour continuous infusion for 5 of 7 days (Monday-Friday) of each RT week for approximately 5 weeks. Patients will continue for full 5.5 weeks unless unacceptable toxicity occurs.

SUMMARY:
This is a Phase 1/ 2, open-label, single-center study of preoperative chemoradiotherapy and AT-101 in patients with locally advanced esophageal or gastroesophageal junction cancer.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients age ≥18 years
* Histologically confirmed primary (non-recurrent) adenocarcinoma (AC) or squamous cell carcinoma of the esophagus or AC of the gastroesophageal (GE) junction.
* For Phase 1: Phase 1 patients must have unresectable disease (Stage II to IVa). A patient can be unresectable for medical reasons or technical reasons but eligible for chemoradiation.
* For Phase 2: Phase 2 patients must have resectable cancer defined as: T2, T3, N0; OR T1-3, N+
* Patients must have archived tumor tissue to correlate tumor biomarker expression with clinical response. Availability of tumor specimens in paraffin blocks or at least two unstained slides must be confirmed prior to study entry. Results will not be used to determine patient eligibility for the study.
* ECOG performance status 0-1
* Adequate hematologic function
* Adequate liver and renal function
* Ability to swallow and retain oral medication.

Exclusion Criteria:

* Patients with distant metastasis, including M1b lymph node status. (M1b status allowed on Phase I only for patients appropriate for chemoradation). Lymph nodes suspicious of M1b status by diagnostic imaging must be verified by fine-needle aspiration cytology. (Phase 2 only)
* For Phase 2: Patients with positive pleural, pericardial, or peritoneal cytology.
* For Phase 2: Patients with carcinoma of the cervical esophagus.
* For Phase 2: Patients with clinical evidence of metastasis to cervical or supraclavicular lymph nodes.
* Prior chemotherapy or radiotherapy for esophageal or gastroesophageal junction cancer. Phase 1 patients with prior chemotherapy are permitted to enter.
* Prior radiotherapy that would overlap the anticipated study treatment fields or radiotherapy to >30% of the marrow cavity (no prior chest irradiation).
* Patients with malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel are excluded. Subjects with ulcerative colitis, inflammatory bowel disease, or partial or complete small bowel obstruction are also excluded.
* Pregnant or nursing females. Fertile patients (male and female) must use effective contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2007-08; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Phase 1: Safety and tolerability of AT-101 in combination with chemoradiotherapy, and determine a dose for Phase 2. Phase 2: Determine the pathologic complete response (pathCR) rate and to correlate tumor biomarker expression with clinical response. | 1 year

SECONDARY OUTCOMES:
To assess the safety and toxicity of chemoradiotherapy and AT-101 in patients with esophageal or gastroesophageal junction cancer. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Lance Leopold, MD, Study Director — Ascenta Therapeutics, Inc.
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States